CLINICAL TRIAL: NCT00893139
Title: A Study of AL-38583 Ophthalmic Solution 0.05%, 0.010% Versus AL-38583 Vehicle for Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-08-077
Record Dates: First submitted 2009-05-04; First posted 2009-05-05 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Dry Eye
Keywords: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AL-38583 0.05% (Experimental): AL-38583 ophthalmic solution 0.05%, 1 drop per eye, 3 times a day, for 35 days
  Interventions: Drug: AL-38583 ophthalmic solution 0.05%
- AL-38583 0.10% (Experimental): AL-38583 ophthalmic solution 0.10%, 1 drop per eye, 3 times a day, for 35 days
  Interventions: Drug: AL-38583 ophthalmic solution 0.10%
- AL-38583 vehicle (Placebo Comparator): Inactive ingredients used as a placebo comparator, 1 drop per eye, 3 times a day, for 35 days
  Interventions: Drug: AL-38583 vehicle

INTERVENTIONS:
Drug: AL-38583 ophthalmic solution 0.05%
  Arms: AL-38583 0.05%
Drug: AL-38583 ophthalmic solution 0.10%
  Arms: AL-38583 0.10%
Drug: AL-38583 vehicle — Inactive ingredients used as a placebo comparator
  Arms: AL-38583 vehicle

SUMMARY:
The purpose of this study is to determine whether AL-38583 ophthalmic solution is effective for treatment of signs and symptoms of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Composite corneal staining score of greater than 5 in one or both eyes.
* Schirmer II score of greater than 4 mm.
* OSDI score of greater than 23.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any medical condition (systemic or ophthalmic) that may, in the opinion of the investigator, preclude the safe administration of the test article or safe participation in this study.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 765 (Actual)
Dates: Start 2009-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in sodium fluorescein corneal staining score | Baseline, up to Day 35

SECONDARY OUTCOMES:
Mean change from baseline in phenol red thread length | Baseline, up to Day 35

CONTACTS AND LOCATIONS:
Overall Officials: Ravaughn Williams, OD, MS, Study Director — Alcon Research